CLINICAL TRIAL: NCT03705143
Title: The Behavioral Activation for Chinese Substance Users (C-BA) Research Protocol
Brief Title: Behavioral Activation for Heroin Use in China: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Wuhan Center for Disease Control and Prevention (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-0885
Record Dates: First submitted 2018-10-02; First posted 2018-10-15 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Substance-Related Disorders; Mood Disorders; Behavioral Activation Treatment; Mental Disorders
Keywords: Disease; Depressive Disorder; Depression; Mood Disorders; Mental Disorders; Substance use Disorders; Chinese heroin user; Culture
MeSH Terms: conditions — Substance-Related Disorders; Mood Disorders; Mental Disorders; Disease; Depressive Disorder; Depression | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (Placebo Comparator): Participants will receive no additional intervention besides the services they are currently receiving at the MMT clinic.
  Interventions: Behavioral: Treatment as usual
- Chinese translated LETS ACT (Experimental): In addition to services participants are currently receiving at the MMT clinic, individuals will attend six group-based one-hour behavioral activation treatment sessions.
  Interventions: Behavioral: Chinese translated LETS ACT

INTERVENTIONS:
Behavioral: Treatment as usual — Treatment as Usual participants will receive the treatment typically provided to patients at the MMT clinic in Wuhan, China.
  Other Names: TAU
  Arms: Treatment as Usual
Behavioral: Chinese translated LETS ACT — The Chinese translated Behavioral Activation (C-BA) will be provided in Mandarin. C-BA treatment includes psychoeducation regarding the link between mood and behavior, identification of values/goals/activities across life areas, planning and tracking of daily value driven activities.
  Other Names: Chinese translated Behavioral Activation
  Arms: Chinese translated LETS ACT

SUMMARY:
This was a single-site two-arm parallel-group trial conducted in a Methadone Maintenance Treatment (MMT) Clinic that provides medication service for 254 heroin users in Wuhan, China. Once consented and completed the pre-treatment assessment, participants were randomized to receive either the Chinese translated behavioral activation treatment for substance use (C-BA) or treatment as usual (TAU). Research assessments occurred at pre-treatment, post-treatment, and 1- and 3-months follow-ups.

The primary purpose of this study is to:

1. Evaluate the feasibility, acceptability, and efficacy of the Chinese-translated behavioral activation treatment for substance use (C-BA), an evidence based intervention developed to address the individual and psychological needs of Chinese substance users.

The secondary purpose of this study is to:

Examine the underlying mechanism of C-BA by studying the relationship between change in substance use related outcomes and associated psychological constructs (e.g. levels of behavioral activation and depression).

DETAILED DESCRIPTION:
Over 83% registered drug users in China are primary heroin users. Heroin use is associated with numerous severe health consequences, including elevated risk for HIV, STDs, and fatal overdose. Methadone maintenance treatment (MMT) has become the standard treatment approach for heroin use that show effectiveness in reducing drug injection, HIV transmission, and criminal activities associated with heroin use in China. Nevertheless, dropout rates among MMT seekers is high in China (50%-70% drop out rate three months post treatment initiation), and research suggests that it is important to provide psychosocial treatments for substance use along with MMT. The combined treatment may both increase treatment adherence and result in superior substance use treatment outcomes.

The Chinese-translated behavioral activation treatment (C-BA) for substance use was translated from the Life Enhancement Treatment for Substance Use (LETS ACT), an evidence based treatment for substance use in the United States. C-BA may fit the need in China because it is a cost-effective and low training-burden treatment designed to be implemented under settings with limited resources. Similar to LETS ACT, C-BA aims to improve substance use outcomes by helping the individuals engage in drug-free value based activities.

Recent studies reported that compared to participants in the supportive counseling group, individuals who received LETS ACT shows significantly higher abstinence rates at 3 months [odds ratio (OR) = 2.2, 95% confidence interval (CI) = 1.3-3.7], 6 months (OR = 2.6, 95% CI= 1.3-5.0) and 12 months (OR = 2.9, 95% CI = 1.3-6.1) post-treatment. Additionally, LETS ACT participants reported significantly fewer adverse consequences from substance use at 12 months post-treatment [B = 4.50, standard error (SE) = 2.17, 95% CI = 0.22-8.78]. In another pilot study, the feasibility and acceptability of C-BA was evaluated among six Chinese international students in the United States. Results suggest that C-BA is associated with both statistical and clinical improvement in depressive symptoms and access to environmental rewards up until 1 month post treatment. The study has a 100% research and treatment retention rate, high homework completion rate (> 80% completion rate), and all participants reported that C-BA is highly culturally acceptable. These preliminary evidence support the feasibility of implementing C-BA among Chinese substance users.

Taken together, research suggests that C-BA could be a feasible treatment that has the potential to reduce substance use, alleviate depressive symptoms, and improve levels of behavioral activation among Chinese heroin users. To date, no study has investigated the feasibility, acceptability and efficacy of C-BA among Chinese heroin users seeking MMT treatment. The present study aims to address this need by conducting a randomized controlled trial to examine the acceptability, feasibility, and efficacy of C-BA among 90 Chinese heroin users seeking MMT. In the current study, the investigators will examine the treatment specifically with regard to major depression, reinforcement, adherence to MMT, and abstinence from substance use. The investigators will also examine the underlying mechanism of C-BA by studying the relationship between change in substance use related outcomes and associated psychological constructs (e.g. levels of behavioral activation and depression).

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving Methadone Maintenance Treatment
* Between 18 and 65
* No outstanding health conditions
* Has received MMT treatment for more than three weeks
* Will continue MMT treatment for at least four more weeks

Exclusion Criteria:

* Reading level below 5th grade
* Psychosis
* PTSD
* The inability to give informed, voluntary, written consent to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
Change in the % substance use days over time | Pretreatment through 3-month post treatment discontinuation
  The frequency of substance use over the past 30 days was measured by a Timeline Followback Interview (TLFB).The % was calculated by using the # of days participants used substance during the 30-day period prior to each assessment point divided by 30. Data was collected at pre-treatment, post-treatment, 1-month post treatment discontinuation and 3-month post treatment discontinuation. The exception is the post-treatment assessment which will only includes a 21 day period.
  The TLFB is a questionnaire in which the subject is asked to self-report types and frequency of substance use for the past 30 days. On the group level, statistical methods such as multi-level modeling (MLM) will be used to assess group differences in change in % of days using substance over the course of the study. On the individual level, statistical methods such as Reliable Change Index (RCI) will be used to assess change in % of days using substance that is clinically significant.

SECONDARY OUTCOMES:
Change in # of participants showing positive urinalysis results over the course of the study | Pretreatment through 3-month post treatment discontinuation
  Urinalysis is a biological measure of substance use. Statistical methods such as multi-level modeling (MLM) will be used to assess group differences in change in # of participants showing positive urinalysis results over time. Data was collected at pre-treatment, post-treatment, 1-month post treatment discontinuation and 3-month post treatment discontinuation.
Change in Beck Depression Inventory-II (BDI-II) Score over the course of the study | Pretreatment through 3-month post treatment discontinuation
  The BDI-II is a 21-item self-report measure of depressive symptoms. Scores range from 0 - 63, with higher scores indicating more severe depressive symptoms. On the group level, statistical methods such as multi-level modeling (MLM) will be used to assess group differences in change in BDI-II total scores over time. On the individual level, statistical methods such as Reliable Change Index (RCI) will be used to assess change in BDI-II total scores that are clinically significant. Data was collected at pre-treatment, post-treatment, 1-month post treatment discontinuation and 3-month post treatment discontinuation.
Change in Behavioral Activation for Depression Scale (BADS) Scores over the course of the study | Pretreatment through 3-month post treatment discontinuation
  The BADS is a 25-item self-report measure of overall level of activity involvement. Scores range from 25 - 175, with higher scores indicating greater levels of activity involvement. On the group level, statistical methods such as multi-level modeling (MLM) will be used to assess group differences in change in BADS total scores over time. On the individual level, statistical methods such as Reliable Change Index (RCI) will be used to assess change in BADS total scores that is clinically significant. Data was collected at pre-treatment, post-treatment, 1-month post treatment discontinuation and 3-month post treatment discontinuation.
Change in Reward Probability Index (RPI) Scores over the course of the study | Pretreatment through 3-month post treatment discontinuation
  The RPI is a 20-item self-report measure used to assess environmental reward and punishment. Scores range from 0 - 60, with higher scores indicating greater levels of access to environmental rewards. On the group level, statistical methods such as multi-level modeling (MLM) will be used to assess group differences in change in RPI total scores over time. On the individual level, statistical methods such as Reliable Change Index (RCI) will be used to assess change in RPI total scores that is clinically significant. Data was collected at pre-treatment, post-treatment, 1-month post treatment discontinuation and 3-month post treatment discontinuation.
Change in % days participants take methadone at the clinic over the course of the study | Pretreatment through 3-month post treatment discontinuation
  Methadone treatment adherence is measured by participant's % of days visiting MMT clinic during the course of the study. On the group level, statistical methods such as multi-level modeling (MLM) will be used to assess group differences in change in % days participants take methadone at the clinic over time. On the individual level, statistical methods such as Reliable Change Index (RCI) will be used to assess change in % days participants take methadone at the clinic that is clinically significant. Data was collected at pre-treatment, post-treatment, 1-month post treatment discontinuation and 3-month post treatment discontinuation.
Change in % days participants engaged in Daily Goals Form over the course of the study | Pretreatment through 3-month post treatment discontinuation
  The Daily Goals Form is used to measure Treatment Engagement. The % days participants engaged in Daily goals Form was calculated by dividing the total # of days participants completed the "Daily Goals Form" by the total # of days they were given the opportunity to complete the "Daily Goals Form." Data was collected at pre-treatment, post-treatment, 1-month post treatment discontinuation and 3-month post treatment discontinuation.
  Once the % is calculated, on the group level, statistical methods such as multi-level modeling (MLM) will be used to assess group differences in change in % days participants engaged in Daily Goals Form over time. On the individual level, statistical methods such as Reliable Change Index (RCI) will be used to assess change in % days participants engaged in Daily Goals Form that is clinically significant.
Feasibility of the treatment | Three weeks since pre-treatment assessment
  Feasibility of the treatment was measured by the following outcomes: % of participated treatment sessions and scores of the Working Alliance Inventory (WAI).
  WAI is a 12-item self-report measure of the quality of therapist-client alliance. Scores range from 12 to 48, with higher scores indicating stronger working alliance.
Acceptability o the treatment | Three weeks since pre-treatment assessment
  Acceptability of the treatment was measured scores of the Treatment Acceptability Questionnaire (TAQ).
  Treatment Acceptability Questionnaire (TAQ) is a 6-item self-report measure of patient's rating of the treatment's acceptability, ethics, effectiveness, negative side effects, therapist knowledge, and therapist trustworthiness. Score range between 6 and 42, with higher scores indicate greater treatment acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Daughters, Ph.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Wuhan Center for Disease Control and Prevention, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daughters SB, Braun AR, Sargeant MN, Reynolds EK, Hopko DR, Blanco C, Lejuez CW. Effectiveness of a brief behavioral treatment for inner-city illicit drug users with elevated depressive symptoms: the life enhancement treatment for substance use (LETS Act!). J Clin Psychiatry. 2008 Jan;69(1):122-9. doi: 10.4088/jcp.v69n0116. PMID 18312046
- [Background] Daughters SB, Magidson JF, Anand D, Seitz-Brown CJ, Chen Y, Baker S. The effect of a behavioral activation treatment for substance use on post-treatment abstinence: a randomized controlled trial. Addiction. 2018 Mar;113(3):535-544. doi: 10.1111/add.14049. Epub 2017 Nov 19. PMID 28963853
- [Background] Daughters, S. B., Magidson, J. F., Lejuez, C. W., & Chen, Y. (2016). LETS ACT: a behavioral activation treatment for substance use and depression. Advances in Dual Diagnosis, 9(2/3), 74-84.
- [Background] Chawarski MC, Zhou W, Schottenfeld RS. Behavioral drug and HIV risk reduction counseling (BDRC) in MMT programs in Wuhan, China: a pilot randomized clinical trial. Drug Alcohol Depend. 2011 Jun 1;115(3):237-9. doi: 10.1016/j.drugalcdep.2010.09.024. Epub 2010 Dec 14. PMID 21159452
- [Background] Wang L, Wang N, Wang L, Li D, Jia M, Gao X, Qu S, Qin Q, Wang Y, Smith K. The 2007 Estimates for People at Risk for and Living With HIV in China: Progress and Challenges. J Acquir Immune Defic Syndr. 2009 Apr 1;50(4):414-8. doi: 10.1097/QAI.0b013e3181958530. PMID 19214116
- [Background] Yin L, Qin G, Ruan Y, Qian HZ, Hao C, Xie L, Chen K, Zhang Y, Xia Y, Wu J, Lai S, Shao Y. Nonfatal overdose among heroin users in southwestern China. Am J Drug Alcohol Abuse. 2007;33(4):505-16. doi: 10.1080/00952990701407223. PMID 17668336
- [Background] Zhang L, Chow EP, Zhuang X, Liang Y, Wang Y, Tang C, Ling L, Tucker JD, Wilson DP. Methadone maintenance treatment participant retention and behavioural effectiveness in China: a systematic review and meta-analysis. PLoS One. 2013 Jul 26;8(7):e68906. doi: 10.1371/journal.pone.0068906. Print 2013. PMID 23922668
- [Background] Feng Y, Wu Z, Detels R, Qin G, Liu L, Wang X, Wang J, Zhang L. HIV/STD prevalence among men who have sex with men in Chengdu, China and associated risk factors for HIV infection. J Acquir Immune Defic Syndr. 2010 Feb;53 Suppl 1(Suppl 1):S74-80. doi: 10.1097/QAI.0b013e3181c7dd16. PMID 20104114
- [Background] Sun HM, Li XY, Chow EP, Li T, Xian Y, Lu YH, Tian T, Zhuang X, Zhang L. Methadone maintenance treatment programme reduces criminal activity and improves social well-being of drug users in China: a systematic review and meta-analysis. BMJ Open. 2015 Jan 8;5(1):e005997. doi: 10.1136/bmjopen-2014-005997. PMID 25573521
- [Background] Marienfeld C, Liu P, Wang X, Schottenfeld R, Zhou W, Chawarski MC. Evaluation of an implementation of methadone maintenance treatment in China. Drug Alcohol Depend. 2015 Dec 1;157:60-7. doi: 10.1016/j.drugalcdep.2015.10.001. Epub 2015 Oct 8. PMID 26601934
- [Background] Lu L, Fang Y, Wang X. Drug abuse in China: past, present and future. Cell Mol Neurobiol. 2008 Jun;28(4):479-90. doi: 10.1007/s10571-007-9225-2. Epub 2007 Nov 8. PMID 17990098